CLINICAL TRIAL: NCT04304417
Title: The Role of Group Identity on the Community Integration of People With Severe Mental Disorder
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Carolina Ugidos Gutiérrez, Principal Investigator, Universidad Complutense de Madrid
Other Study IDs: 2019/20-020
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Bipolar Disorder; Personality Disorders; Psychotic Disorders
Keywords: Severe Mental Disorder; Community Integration; Group Identity; Stigma; Dehumanization
MeSH Terms: conditions — Bipolar Disorder; Personality Disorders; Psychotic Disorders; Mental Disorders; Social Stigma; Dehumanization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study analyzes which variables enhance or hinder community integration among people with severe mental disorder. Participants will complete a questionnaire to test our hypotheses:

* Hypothesis 1: group identification predicts less self-dehumanization and self-stigma, and more empowerment, these in turn predict more community integration.
* Hypothesis 2: the relationship between group identification and self-dehumanization and self-stigma is moderated by group value.
* Hypothesis 3: when group identification is low, group identification predicts higher community integration, but this relationship is mediated by diagnosis concealment.

DETAILED DESCRIPTION:
Community integration, which includes physical integration (e.g. participation in activities, as well as use of goods and services in the community in a self-initiated manner), social integration (e.g. quantity and quality of social relationships) and psychological integration (e.g. perception of belongingness to the community), is a necessary element to achieve personal recovery among people with severe mental disorder (SMD).

Group identification, based on Social Identity Theory, emphasizes an individual's definition of who they are in relation to their group membership. When individuals have a strong tendency to define their self-concept in terms of the group they belong to and uphold the values of their group, they are said to have high identification with the group. Group value, on the other hand, refers to the evaluative judgment of one's social group, which reflects the extent to which individuals feel positively or negatively toward their ingroup, and people who have positive perceptions toward their group are more strongly identified with it.

Self-dehumanization is the process by which people dehumanize themselves. This can happen in two ways: when they perceiving themselves as unintelligent, amoral, irrational, wild, etc.; thus perceived as animal-like, it is called animalistic dehumanization; or when they perceive themselves as lacking emotion, warmth, vitality, etc.; perceived as object-like, which is referred to as mechanistic dehumanization.

Self-stigma occurs when people accept the negative stereotypes about their in-group apply to themselves. This has shown to influence the community integration of people with SMD.

Empowerment is understood as the process by which people, organizations and communities acquire control over their own lives. People with SMD who endorsed higher group value were more likely to be involved in educating the public about mental health and helping others with mental disorder, which are considered a behavioral manifestation of empowerment.

In order to test the hypotheses previously mentioned, the users of the public centers of social care for people with SMD of the State of Madrid (Spain) will be contacted. The inclusion criteria are: to have a diagnosis of SMD and disorder consciousness. The exclusion criteria are: to be underage and legally incapacitated. Participants will complete a pencil-and-paper questionnaire, including the measurement of the variables previously mentioned and some socio-demographical questions, in the centers they attend.

The analytical program SPSS.25 (Statistical Package for the Social Sciences) will be used to conduct the appropriate test of hypothesis (correlation, regression, mediation, moderation).

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of severe mental disorder.
* Having disorder consciousness.

Exclusion Criteria:

* Being underage.
* Being legally incapacitated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study are adult people with a diagnosis of severe mental disorder (SMD), who are users of the public centers of social care for people with SMD of the State of Madrid in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Physical integration | 1 day. Measured the day of the study.
  Self-reported frequency of activities realized outdoors, measured with the subscale 'Leisure and community' from the 'Independent living skills survey'. Each item is scored from 1 (never) to 5 (always).
Social integration | 1 day. Measured the day of the study.
  Self-reported frequency of support available, measured with the Medical Outcome Study Social Support Survey (MOS-SSS). Each item is scored from 1 (never) to 5 (always).
Psychological integration | 1 day. Measured the day of the study.
  Self-reported feeling of belonging to the general community and to the community of people with mental disorder. It is measured with the subscale 'Belonging' from the 'Community Integration Measure'. Each item is scored from 1 (I totally disagree) to 5 (I totally agree).

SECONDARY OUTCOMES:
Self-dehumanization | 1 day. Measured the day of the study.
  Haslam's scale of Human Nature and Human Uniqueness to measure wether participants think different adjectives describe them. Each item is scored from 1 (I am not at all like that) to 7 (I am exactly like that).
Self-stigma | 1 day. Measured the day of the study.
  Self-reported measure of participants' internalized stigma using the 'Internalized Stigma of Mental Illness Inventory-9'. Each item range from 1 (I totally disagree) to 4 (I totally agree).
Empowerment | 1 day. Measured the day of the study.
  Self-reported measure of empowerment using the subscales 'Self-esteem-self-efficacy' and 'Community activism and autonomy' from the empowerment scale developed by Rogers, Chamberlin, Ellison y Crean (1997), and the subscale 'disclosure' developed by King et al. (2007). Items range from 1 (I totally disagree) to 4 (I totally agree).
Group identity | 1 day. Measured the day of the study.
  The subscales 'Interconnection of self with the group' and 'Sense of interdependence' from the team identity scale developed by Heere and James (2007). Items range from 1 (I totally disagree) to 7 (I totally agree).
Group value | 1 day. Measured the day of the study.
  The subscale 'Private evaluation' from the team identity scale developed by Heere and James (2007). Items range from 1 (I totally disagree) to 7 (I totally agree).

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Ugidos, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Grupo 5, Madrid, State of Madrid, Spain

IPD SHARING:
Plan to Share IPD: No